CLINICAL TRIAL: NCT04118348
Title: Evaluating the Efficacy of Different Electronic Medical Record Alerts to Increase Pediatric Lipid Screening Across a Large Integrated Health System
Brief Title: Evaluating the Efficacy of Pediatric Lipid Screening Alerts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Screening
Other Study IDs: 2019-0418
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Hypercholesterolemia; Hypercholesterolemia, Familial; Hypercholesteremia in Children; Hyperlipidemia in Children
Keywords: Optimal default; Best practice alert; Health maintenance topic
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Passive Control (No Intervention): Will consist of no alerts and will serve to examine lipid panel screening rates given the current standard of care. After 6 months, providers in this (and other conditions) will receive the alert(s) with the best demonstrated success in increasing screening rates.
- Best Practice Alert (BPA-only) (Experimental): Will consist of a BPA that fires for providers during a visit with an eligible 9-11 year-old patient. This is an active opt-in alert wherein the provider must respond, either confirming the prescription of a lipid panel or opting out with an acknowledgment/reason for declining the test. The BPA will include a recommendation to administer the screen in combination with existing scheduled bloodwork.
  Interventions: Behavioral: Best Practice Alert
- Health Maintenance Topic (HMT-only) (Experimental): Will consist of an HMT in Epic that is present for providers at their visit with an eligible patient. The HMT will be highlighted for enhanced visibility, until or unless action is taken.
  Interventions: Behavioral: Health Maintenance Topic
- BPA+HMT (Experimental): Will consist of both the BPA and HMT presented simultaneously in Epic.
  Interventions: Behavioral: Best Practice Alert; Behavioral: Health Maintenance Topic

INTERVENTIONS:
Behavioral: Best Practice Alert — An Epic screen pops up for a provider during an eligible 9-11 year-old patient's visit. A prompt requires that the provider respond, either confirming the prescription of a lipid panel or opting out with an acknowledgment/reason for declining the test.
  Arms: BPA+HMT; Best Practice Alert (BPA-only)
Behavioral: Health Maintenance Topic — An Epic health maintenance topic appears for a provider during an eligible 9-11 year-old patient's visit. The HMT will be highlighted for enhanced visibility, until or unless action is taken.
  Arms: BPA+HMT; Health Maintenance Topic (HMT-only)

SUMMARY:
The purpose of the study is to evaluate prospectively the impact of different system alerts on the prescription of lipid panels to pediatric Geisinger patients (9-11 years old), as per the now-universal guidelines. This will help quantify the relative effectiveness of different alerts and combinations of alerts on provider prescribing behavior and patient uptake of screening.

DETAILED DESCRIPTION:
Patients who are eligible for this study will be randomized into one of four groups via an Epic electronic medical record (EMR) randomization algorithm run automatically at the time of the visit:

1. Control group (6-month delay before their providers will receive an alert)
2. Health maintenance topic (HMT)
3. Best practice alert (BPA)
4. Best practice alert and health maintenance topic (BPA+HMT)

Geisinger Health System will introduce Epic's Storyboard panel (a novel way of summarizing patient information in the EMR) approximately one month into this study. The analysis plan will therefore test for the potential impact of this change.

The providers will be prompted to discuss and order screening lipid study that is non fasting at the time of the visit with the patient, based on the alerts above. Some families will have an alert in their MyGeisinger portal stating that a health maintenance test is due and to discuss with their provider.

Outcomes will be reviewed and classified as followed,

Outcomes will include lipid screening orders by providers (yes/no) and screening completions by patients (yes/no). The following descriptive results will also be provided:

1. Lipid screening ordered
2. Lipid screening ordered and completed
3. Lipid screening ordered but not completed
4. Lipid screening declined with reason why
5. Alert not acted on at all

Analysis will account for the nesting of patients within providers; this will include provider as a random effects variable in a series of multilevel binomial logistic regression models, to account for potential correlation with patients. If the intraclass correlation coefficient is low, only the patient-level logistic regression models will be conducted. In the first model, the passive control will serve as the reference group, to test whether each of the active alert conditions have a significant impact on the outcomes. In the second model, the BPA-only condition will serve as the reference group, to test whether HMT and BPA+HMT offer significant improvements in performance. Finally, the third model will use the HMT-only condition as the reference, to test whether BPA+HMT has a significantly greater impact on the outcomes. Storyboard X Condition interactions will be tested within the models, and if any are significant, the series of models will be conducted separately on patients prior to, and after, implementation of Storyboard in Epic, to test whether and how results replicate in the different contexts.

ELIGIBILITY:
Inclusion criteria:

* male or female patients between the ages of 9 - 11
* seen within a primary care, cardiology, endocrinology, urgent care (CareWorks), or nutrition clinic at Geisinger

Exclusion criteria:

* patients who have completed a lipid screen in the EMR
* patients who were determined to have familial hypercholesterolemia based on prior screening

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13340 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-10-11 (Actual); Study Completion 2020-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

REFERENCES:
- [Derived] Goren A, Santos HC, Davis TW, Lowe RB, Monfette M, Meyer MN, Chabris CF. Comparison of Clinical Decision Support Tools to Improve Pediatric Lipid Screening. J Pediatr. 2024 Jun;269:113973. doi: 10.1016/j.jpeds.2024.113973. Epub 2024 Feb 22. PMID 38401785

RESULTS

PARTICIPANT FLOW:
Groups:
- Best Practice Alert (BPA-only): Will consist of a BPA that fires for providers during a visit with an eligible 9-11 year-old patient. This is an active opt-in alert wherein the provider must respond, either confirming the prescription of a lipid panel or opting out with an acknowledgment/reason for declining the test. The BPA will include a recommendation to administer the screen in combination with existing scheduled bloodwork.
  When referring to study arms, BPA refers to participants who triggered BPAs only.
- Health Maintenance Topic (HMT-only): Will consist of an HMT in Epic that is present for providers at their visit with an eligible patient. The HMT will be highlighted for enhanced visibility, until or unless action is taken.
  When referring to study arms, HMT refers to participants who triggered HMTs only.
- BPA+HMT: Will consist of both the BPA and HMT presented simultaneously in Epic. This is a separate group of participants compared to the BPA-only and HMT-only arms.
  When referring to study arms, BPA+HMT refers to participants who triggered a combination of BPA and HMT.
Period: Overall Study
Arm/Group | Passive Control | Best Practice Alert (BPA-only) | Health Maintenance Topic (HMT-only) | BPA+HMT
Started | 3416 | 3265 | 3441 | 3218
Completed (Random assignment happened at the patient encounter) | 3416 | 3265 | 3441 | 3218
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only data related to test orders was pulled for this analysis. No demographic or other baseline data were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Passive Control | Best Practice Alert (BPA-only) | Health Maintenance Topic (HMT-only) | BPA+HMT | Total
Number analyzed (Participants) | 3416 | 3265 | 3441 | 3218 | 13340
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3416 | 3265 | 3441 | 3218 | 13340
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3416 | 3265 | 3441 | 3218 | 13340

OUTCOME MEASURES:

1. Primary Outcome: Lipid Panel Order
Description: Provider ordered a lipid panel to an eligible patient during the patient's first visit within the study period (binary variable).
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Control | Best Practice Alert (BPA-only) | Health Maintenance Topic (HMT-only) | BPA+HMT
Number analyzed (Participants) | 3416 | 3265 | 3441 | 3218
Participants | 156 | 454 | 236 | 494
Statistical Analysis 1: Comparison: Passive Control vs BPA+HMT; Passive control was set as the reference group; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 5.73, 95% CI 2-sided [4.46 to 7.36] — BPA+HMT is the numerator
Statistical Analysis 2: Comparison: Passive Control vs Best Practice Alert (BPA-only); Passive control was set as the reference group; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 4.87, 95% CI 2-sided [3.79 to 6.27] — BPA-only is the numerator
Statistical Analysis 3: Comparison: Passive Control vs Health Maintenance Topic (HMT-only); Passive control was set as the reference group; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.28 to 2.19] — HMT-only is the numerator
Statistical Analysis 4: Comparison: Health Maintenance Topic (HMT-only) vs BPA+HMT; HMT was set as the reference group; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 3.43, 95% CI 2-sided [2.73 to 4.29] — BPA+HMT is the numerator
Statistical Analysis 5: Comparison: Best Practice Alert (BPA-only) vs Health Maintenance Topic (HMT-only); HMT was set as the reference group; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 2.92, 95% CI 2-sided [2.32 to 3.66] — BPA-only is the numerator
Statistical Analysis 6: Comparison: Best Practice Alert (BPA-only) vs BPA+HMT; BPA was set as the reference group; Test type: Superiority; p = .114, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.96 to 1.43] — BPA+HMT is the numerator

2. Primary Outcome: Lipid Panel Screening
Description: Patient completed a lipid panel screening within seven days of the patient's first visit (binary variable). This screening is not linked to any order made at the patient's first visit (i.e., Outcome Measure 1).
Time Frame: 1 week
Population: We examined all completions made during the time frame, regardless of an order being made at their initial visit. This outcome measure thus covers completions from orders made during the first or any subsequent visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Passive Control | Best Practice Alert (BPA-only) | Health Maintenance Topic (HMT-only) | BPA+HMT
Number analyzed (Participants) | 3416 | 3265 | 3441 | 3265
Participants | 47 | 98 | 70 | 120
Statistical Analysis 1: Comparison: Passive Control vs BPA+HMT; Passive control was set as the reference group; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 2.90, 95% CI 2-sided [2.02 to 4.15] — BPA+HMT is the numerator
Statistical Analysis 2: Comparison: Passive Control vs Best Practice Alert (BPA-only); Passive control was set as the reference group; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 2.28, 95% CI 2-sided [1.57 to 3.30] — BPA-only is the numerator
Statistical Analysis 3: Comparison: Passive Control vs Health Maintenance Topic (HMT-only); Passive control was set as the reference group; Test type: Superiority; p = .030, Regression, Logistic; Odds Ratio (OR) = 1.54, 95% CI 2-sided [1.04 to 2.27] — HMT-only is the numerator
Statistical Analysis 4: Comparison: Health Maintenance Topic (HMT-only) vs BPA+HMT; HMT was set as the reference group; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.37 to 2.59] — BPA+HMT is the numerator
Statistical Analysis 5: Comparison: Best Practice Alert (BPA-only) vs Health Maintenance Topic (HMT-only); HMT was set as the reference group; Test type: Superiority; p = .021, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.06 to 2.06] — BPA-only is the numerator
Statistical Analysis 6: Comparison: Best Practice Alert (BPA-only) vs BPA+HMT; BPA was set as the reference group; Test type: Superiority; p = .107, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.95 to 1.71] — BPA+HMT is the numerator

ADVERSE EVENTS:
Time Frame: We did not report a time frame as we did not actively collect adverse event data.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed. No adverse events were evaluated, as only data from orders and completed tests were gathered. Mortality was not a risk associated with participation in our study.
Arm/Group | Passive Control | Best Practice Alert (BPA-only) | Health Maintenance Topic (HMT-only) | BPA+HMT
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The description of the outcome measures was revised to be more accurate. The analysis plan was also modified from the plan outlined in the study description to include corrections for multiple comparisons (i.e., Tukey correction).

Due to limited data access, only information about the orders and completions were given to the researchers. As a result, demographic data and data on adverse effects were not gathered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT04118348/Prot_001.pdf
  • Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT04118348/SAP_003.pdf